CLINICAL TRIAL: NCT05252286
Title: Comparison of Three Types of Bedside Exercise Programs on Physical Functions of Hospitalized Patients
Brief Title: Exercise Strategies for Bedside Cases During Hospitalization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Jia-Ching Chen, Associate professor, Department of physical therapy, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB110-193-A
Record Dates: First submitted 2022-01-22; First posted 2022-02-23 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Disability Physical; Hospitalization
Keywords: Hospital-Associated Disability; self-exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- video watching (Experimental): In the video-watching group, a patient will follow the exercise instructions from watching the video. The exercise content in video are set during the patient conducting the rehabilitation program. Then, the therapist will select 3 to 5 groups of movements pattern needed to be enhanced catching from the video for the patient to practice when returning the bedside after the rehabilitation programs.
  Interventions: Other: video watching
- paper sheet (Active Comparator): For the paper sheet group, the therapist will prepare the exercise leaflet, suitable for the patients, in advance, and select three to five groups of movement exercises on the leaflet that his/her therapist deem the patients needed to be enhanced. When the patients ends his/her rehabilitation program, they can practice following the instructions on the leaflet for them-self in bedside.
  Interventions: Other: paper group
- oral health education group (Placebo Comparator): In the oral health education group, the program is similar to the paper sheet group without providing any exercise paper sheet the patient but oral education.
  Interventions: Other: oral education group

INTERVENTIONS:
Other: video watching — Watching video In this group, when the patient conducts their rehabilitation exercise, the therapist would record the poor physical movement pattern from his/her performance by using the mobile phone or tablet. The patients will be provided with watching video exercise, containing 3-5 items of "their poor physical performance", selected by the therapist as a feedback to let the patient practice when they return their bedside ward after their rehabilitation time. The content of video-watching exercise program will be changed or modified once weekly as the patient improve the physical movement performance.
  Arms: video watching
Other: paper group — In the paper sheet group, the therapist will give three to five poor movement patterns, selected from the patient conducting their rehabilitation program, to practice when returning bedside ward.
  Arms: paper sheet
Other: oral education group — the patient only receives the oral exercise education about how to improve their physical performance during their hospital stay.
  Arms: oral health education group

SUMMARY:
Patients after hospital admission would experience the functional decline, so-called Hospital-Associated Disability. This condition could not only impact the patient health function but pose a burden on the family, even more consuming of medical resource in the country. Therefore, in addition to routine rehabilitation program, various bedside exercise programs are provided as an adjunct therapy to prevent functional declination and improve physical mobility for a patient after hospital admission. The aims of the study are conducted to compare the effect of three various bedside exercise programs (exercise based on watching video, oral education and paper sheet) on physical mobility among the hospitalized patients.

This is single-blind randomized control study and patients recruited from Tzu-Chi medical center in eastern Taiwan are ranged from 30 to 90 years old. All participants are randomly assigned to three groups (watching video, oral education and paper sheet). Patients in watching video group are provided with theirs 3 to 5 poor physical performance video recorded on the tablet or mobile phone during the rehabilitation program. The other two groups are provided oral education and paper sheet exercise program, respectively. All three groups patients conduct their bedside exercise programs when they return their ward.

Physical performance tests are evaluated before the intervention and one or two days before discharge by a physical therapist blinded the groups of patient .

ELIGIBILITY:
Inclusion Criteria:

1. Functional dependence evaluated by Barthel Index
2. Patients needed to rehabilitation program referred by medical doctor during hospitalization
3. Be able to follow command and assessment

Exclusion Criteria:

1. Impaired cognition
2. Psychological problem from medical diagnosis
3. Having a potential cardiac risk or severe disease diagnosis from medical doctor

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Barthel Index (BI) | Up to four weeks
  The investigators will use the BI as the primary outcome measure in this study to evaluate activity of daily living at baseline before intervention, one week after intervention, and the time at discharge. BI is scored 0 to 100, the higher score and the better functional performance.

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | four weeks
  The investigators will use the SPPB as the secondary outcome measure in this study to evaluate the lower extremity functioning and physical mobility at baseline before intervention, one week after intervention, and the time at discharge. SPPB is scored 0 to 12, the higher score and the better physical mobility.
Time Up and Go (TUG) | Up to four weeks
  The investigators will use the TUG as the secondary outcome measure in this study to evaluate the balance mobility at baseline before intervention, one week after intervention, and the time at discharge. TUG is recorded as the seconds, the shorter timing and the better balance function.
de Morton Mobility Index (DEMMI) | Up to four weeks
  The investigators will use the DEMMI as the secondary outcome measure in this study to evaluate the physical mobility at baseline before intervention, one week after intervention, and the time at discharge. The DEMMI consists of 15 items with score 0-100, and the higher score, the better performane.
Hand-held dynamometer | Up to four weeks
  The investigators will use the hand-held dynamometer as the secondary outcome measure in this study to evaluate the muscle strength at baseline before intervention, one week after intervention, and the time at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Ching Chen, Principal Investigator — Department of physical therapy, Tzu Chi University
Locations (1):
- Tzu Chi Buddhist General Hospital, Hualien City, Taiwan